CLINICAL TRIAL: NCT02341963
Title: A Prospective, Open-Label Pilot Clinical Trial of Oral Ketamine for Acute Pain Management After Amputation Surgery
Brief Title: A Pilot Clinical Trial of Oral Ketamine for Acute Pain Management After Amputation Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Professor, Department of Anesthesiology, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORA#: 14071504
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Acute Pain Management; Analgesic, Nonopioid; Amputation of Lower Extremity, All Causes
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Ketamine (Experimental): Subjects will receive Oral Ketamine (1.0 mg/kg) ) presurgery and 3 days postsurgery (including surgery day).
  Interventions: Drug: Oral Ketamine

INTERVENTIONS:
Drug: Oral Ketamine — Oral ketamine (Ketamine HCL injection, 100 mg/ml, USP, Hospira)

SUMMARY:
The purpose of this pilot study is to test the safety of oral ketamine to treat acute pain after amputation surgery. The objective of the proposed research is to conclusively determine if oral ketamine is a safe alternative analgesic to opioid for acute pain in subjects undergoing elective amputation of the lower extremity. All participants will receive oral ketamine.

DETAILED DESCRIPTION:
A prospective open-label clinical trial to decrease the incidence of expected side effects of oral ketamine dose administered presurgery and postsurgery, in 10 subjects undergoing elective amputation of the lower extremity. The primary outcome measure is the incidence of adverse events. Secondary outcome measures are decreased acute pain levels and decreased incidence of stump and phantom limb pain at 6 months. Enrollment of participants will occur at Rush University Medical Center (Rush), Chicago, Illinois. Consented participants will be included in the study undergoing elective amputation of the lower extremity from all causes.

Rationale for using oral ketamine for acute pain after amputation surgery:

The common analgesic, morphine, has a narrow therapeutic window and numerous side effects.1 Ketamine, is a chemically stable compound, non-opioid with analgesic properties at low doses. In addition, ketamine stimulates the cardio-respiratory system which is of great benefit in injured patients.2-4 Ketamine is generally administered by the intravenous (IV) route and provides analgesia via antagonism of the N-Methyl-D-Asparate (NMDA) receptor. Ketamine has the added benefit of a wide therapeutic safety index. IV ketamine has been shown to provide postoperative analgesia in many clinical trials; in particular to reduce opioid consumption.5 Severe acute pain has been shown to progress to chronic pain due to central sensitization.6 Perioperative IV ketamine has been shown in limited studies to decrease the incidence of chronic pain after surgery. However, the IV route of administration of ketamine has limitations due to difficulties with IV placement in certain tactical situations. Therefore, the use of oral ketamine (non-opioid) for the purpose of acute pain management after trauma or surgery is highly desirable.

Pharmacokinetic studies: Oral ketamine may seem disadvantageous because of 17% bioavailability, mainly due to first-pass drug metabolism in the liver. However, there is not a wide variability in bioavailability from patient-to-patient (mean 16.6%, Standard Error (SE) = 2.8%) and hence a predictable oral dosing can be achieved. Although investigators have tested formulations with sublingual or buccal transmucosal administration of ketamine, in practice they fail to increase the ketamine bioavailability versus oral ketamine. Ketamine as nasal spray is problematic for acute use, since the amount of drug is difficult to control using an atomizer.

Day 1 (day of surgery) Before Surgery: An analgesic dose of the oral ketamine (1.0 mg/kg) will be administered one hour before surgery in the preoperative holding area.

If the subject is experiencing any adverse events (e.g. hallucinations) from the 1.0 mg/kg pre-surgery dose of ketamine, then any further ketamine dosing will be delayed until the following day (Day 2). In addition, subsequent subjects will receive a 33% reduction of the pre-surgery dose (i.e. 0.67 mg/kg).

After Surgery: In the recovery room, when subjects are able to swallow, and if there were no adverse events from the pre-surgery ketamine dose, oral ketamine (1.0 mg/kg) will be administered (but no earlier than 8 hours after the pre-surgery dose). No doses will be administered after midnight.

If adverse events have not resolved by the next morning (Day 2), then oral ketamine will be discontinued. In addition, subsequent subjects will receive a 33% reduction in the recovery room dose and/or the last dose of Day 1.

Day 2 (first post-op day) Subjects will receive oral ketamine (1.0 mg/kg) 3 times/day. The first dose will be administered at 6 AM .If a subject experiences any adverse events after the first dose, but one that resolves within 8 hours after that dose, the second dose will be reduced by 33% (1.0 mg/mg to 0.67 mg/kg). If a subject experiences any adverse events after the second dose, but one that resolves within 8 hours, the dose will be reduced again by 33% (0.67 mg/kg to 0.45 mg/kg). If this dose reduction protocol does not eliminate adverse events, then oral ketamine will be discontinued. In addition, subsequent subjects will receive a 33% reduction in the Day 2 oral ketamine doses

Day 3 (second post-op day) (Tapering Down Period) Subjects will receive oral ketamine at half of the previous day final dose (0.5 mg/kg if no dose reductions have occurred), 3 times a day. For example, if the subjects' dose is already at 0.45 mg/kg from the previous day reductions, then the third day dose will be 0.23 mg/kg. The first dose will be administered at 6 AM. Even on the third day if there are adverse events after any dose, but one that resolves within 8 hours after that dose, we will continue to reduce the dose by 33%. If this dose reduction protocol does not eliminate adverse events, then the subject will not receive any more ketamine. In addition, subsequent subjects will receive a 33% reduction in the Day 3 oral ketamine doses.

While in the hospital for 3 days, should breakthrough pain occur, all subjects will receive standard of care pain control medication. All subjects will be discharged according to standard discharge protocol.

Anticipated Adverse Events If a subject experiences adverse events, subjects will be closely monitored every hour until the event resolves. Adverse event duration and resolution time will be recorded. If the adverse event resolves, the next scheduled dose will be reduced by 33%. Each adverse event will be assessed by the Principal Investigator and a clinical relevance determination will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of at least 18 years of age, but not older than 80 years
2. Due to undergo elective major amputation of the lower extremity (above the knee amputation (AKA), below the knee amputation (BKA), total knee amputation (TKA), transmetatarsal amputation (TMA), toe amputation) from all causes.

Exclusion Criteria:

1. Pregnancy
2. Increased intracranial pressure or intraocular pressure
3. Allergy to ketamine
4. Morbid obesity (BMI > 40 kg/m2)
5. Significant comorbidity (ASA physical status classification > 3)
6. Inability to communicate with the investigators
7. Any history of known or suspected drug or alcohol abuse
8. History of impaired liver function
9. Significant history of hallucinations, delusions or other psychiatric medical condition the investigator feels will prevent assessment of adverse events of study drug.
10. Significant psychiatric history; a diagnosis of schizophrenia, bipolar disorder, or severe depression.
11. Exposure to cytochrome P450 3A4 inhibitors or inducers (including grapefruit products) within 2 weeks before enrollment; the inability to avoid these products during ketamine administration.
12. Poorly-controlled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to 72 hours post-surgery or until discharge
  Incidence of adverse events with oral ketamine

SECONDARY OUTCOMES:
Acute Postoperative Pain (NRS (numerical rating scale, 0=no pain, 10=worst imaginable pain) score) | 0 to 72 hours post-surgery
  Patient NRS (numerical rating scale, 0=no pain, 10=worst imaginable pain) score of postoperative pain adjacent to body part that was amputated, at 48 hours post-surgery (average pain over previous 4 h).
Chronic Postoperative Pain (SF-MPQ scale for phantom limb and stump pain;Defense and Veterans Pain Rating Scale (DVPRS) | 1, 3, 6 months post-surgery
  Assessment of stump pain and phantom limb pain using; SF-MPQ scale for phantom limb and stump pain;Defense and Veterans Pain Rating Scale (DVPRS); S-LANSS neuropathic pain scale, RAND 36 Item Health Survey (SF-36) quality of life scale
Pharmacokinetics of Plasma Ketamine and Norketamine Levels (ng/mL) | Post-operative day 1 and 1 and hours after the first morning study drug dose
  The purpose is to be able to relate plasma drug levels to adverse events and side effects.
Liver Function Test | 1 month after surgery and every month until liver function levels return to normal

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, M.D., Principal Investigator — Professor Anesthesiology, Rush Unviersity Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Buvanendran A, Kroin JS, Rajagopal A, Robison SJ, Moric M, Tuman KJ. Oral Ketamine for Acute Pain Management After Amputation Surgery. Pain Med. 2018 Jun 1;19(6):1265-1270. doi: 10.1093/pm/pnx229. PMID 29025089